CLINICAL TRIAL: NCT02194088
Title: Potential for Improved Analgesia From Combined Medication for Superficial Pain
Brief Title: Combined Medication for Improved Analgesia in Superficial Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Robert Edwards, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P001857
Record Dates: First submitted 2013-12-11; First posted 2014-07-18 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac; Acetaminophen; Drug Combinations; Drug Evaluation; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain medication: diclofenac and atropine (Experimental): Diclofenac and Atropine combination drug Provided PO. This is a novel combination. Diclofenac 100mg + Atropine 1.2 mg in one single dose
  Interventions: Drug: Diclofenac and Atropine combination drug
- placebo (Placebo Comparator): Placebo capsules will be delivered in same number as the medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac and Atropine combination drug — Diclofenac will be associated with a small dose of atropine 1.2mg
  Other Names: Analgesic drug; Combination drug; Test drug; Diclofenac and atropine; Atropine and diclofenac
  Arms: Pain medication: diclofenac and atropine
Drug: Placebo — For each capsule of active medication, a capsule of placebo will be provided, identical looking.
  Other Names: Placebo control for the active medication
  Arms: placebo

SUMMARY:
This research study is being done to assess if a combination of medications can enhance the relief of superficial pain (pain at the surface of the skin, such as sunburn pain). The investigators also want to find out if certain genes may be linked to individual differences in experienced efficacy of pain killers. The combination of medications under investigation is diclofenac and atropine. Diclofenac has been approved by the U.S. Food and Drug Administration (FDA) to treat pain. Atropine has been approved by the FDA to treat certain types of poisoning, heartbeat problems, and other diseases but atropine is not approved to treat pain. However, atropine has been used for many years in different European countries to treat painful conditions such as stomach cramps.This research study will compare diclofenac and atropine to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers.
* 18-40 years of age.
* Ability to read and understand English; English can be a second language provided that the participant feels that he/she understand all the questions used in the assessment measures.

Exclusion Criteria:

* Chronic pain condition or chronic or current treatment with any pain medication.
* Presence of any illness or medication use that is judged to interfere with the trial. For example: psychiatric disorder, medication that can influence cognition or emotional processing, i.e. sleep medication, antidepressants, anti-convulsants or opioids.
* Unwillingness to receive brief pain stimulation administered by a heat probe on the hand.
* Allergy or contra-indication to receiving nonsteroidal anti-inflammatory medication and atropine (Treatment with antidepressants, neuroleptics, antihistaminic, levodopa, anti-acids. Pregnancy, breast-feeding, myasthenia gravis, pyloric stenosis, gastro-esophageal reflux, gastric ulcer, constipation, prostatic enlargement, glaucoma, cardio-pulmonary condition -including tachycardia, arrhythmia, arteriosclerosis-, hyperthyroidism, high blood pressure, genetic disease, kidney failure)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Edwards, PHD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berna C, Kirsch I, Zion SR, Lee YC, Jensen KB, Sadler P, Kaptchuk TJ, Edwards RR. Side effects can enhance treatment response through expectancy effects: an experimental analgesic randomized controlled trial. Pain. 2017 Jun;158(6):1014-1020. doi: 10.1097/j.pain.0000000000000870. PMID 28178072
- [Derived] Laursen DR, Nejstgaard CH, Bjorkedal E, Frost AD, Hansen MR, Paludan-Muller AS, Prosenz J, Werner CP, Hrobjartsson A. Impact of active placebo controls on estimated drug effects in randomised trials: a systematic review of trials with both active placebo and standard placebo. Cochrane Database Syst Rev. 2023 Mar 6;3(3):MR000055. doi: 10.1002/14651858.MR000055.pub2. PMID 36877132

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Medication: Diclofenac and Atropine | Placebo
Started | 75 | 25
Completed | 75 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Medication: Diclofenac and Atropine | Placebo | Total
Number analyzed (Participants) | 75 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 25 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.04 (4.75) | 23.16 (3.94) | 23.82 (4.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 14 | 51
  Male | 38 | 11 | 49
Region of Enrollment [Number; unit: participants]
  United States | 75 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores on Standardized Experimental Pain Testing
Description: Pain scores on standardized experimental pain testing, with collection of Visual analog scales (VAS) on a 0-100 scale 0 (no pain)- 100 (worst pain imaginable) Higher values represent a worse outcome (more pain)
Time Frame: baseline and 1 hour pain measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Medication: Diclofenac and Atropine | Placebo
Number analyzed (Participants) | 75 | 25
units on a scale
  Baseline | 59.6 (13.9) | 54.0 (13.9)
  1 hour Assessment | 44.1 (22.7) | 45.3 (18.0)

2. Secondary Outcome: Catechol-O-methyltransferase (COMT) Polymorphism Correlation With Pain Relief
Description: Difference in the baseline pain measurements compared to the 1-hour outcome measure will be correlated with Catechol-O-methyltransferase polymorphism
Time Frame: baseline and 1 hour pain measurement
Population: Data were not collected
Arm/Group | Pain Medication:Diclofenac an Atropine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Side Effects
Description: The investigators aimed assess if these would be a reason for discontinuation of treatment in a population with mild to moderate pain.Side effects will be assessed with a dichotomous measurement (yes/no)
Time Frame: baseline and 1 hour pain measurement
Population: Participants were analyzed in terms of whether they endorsed or not the side effects (yes/no) Participants were not analyzed in terms of severity degree
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Medication: Diclofenac and Atropine | Placebo
Number analyzed (Participants) | 75 | 25
Participants
  Dry mouth | 28 | 7
  Other Side Effects | 4 | 2
  No side effects | 43 | 16

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Pain Medication: Diclofenac and Atropine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/25
Other Adverse Events (participants affected / at risk) | 0/75 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No